CLINICAL TRIAL: NCT01137266
Title: Effects of Transcutaneous Electrical Nerve Stimulation on Pain and Disability in Patients With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Collaborators: Philips Electronics Nederland BV (Industry)
Responsible Party: A. Kolen, Philips Research Eindhoven
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NL2073208008
Record Dates: First submitted 2010-01-28; First posted 2010-06-04 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis
Keywords: chronic pain osteo-arthritis in one or both knees, adults
MeSH Terms: conditions — Osteoarthritis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- skin resistence (Active Comparator): 1) the location with the lowest resistance
  Interventions: Device: TENS
- irradiation (Active Comparator): 2) the site that causes an irradiation sensation
  Interventions: Device: TENS
- random (Active Comparator): 3) a random stimulation site.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — TENS

SUMMARY:
The purpose of this study is to determine the effects of transcutaneous electrical nerve stimulation (TENS) on pain and mobility by comparing different stimulation sitesP:

1. the location with the lowest resistance
2. the location that causes an irradiation sensation
3. a random stimulation site (but within a 10x10cm area of the irradiation site). The effect is defined as the pain VAS baseline-measurement before treatment minus the pain VAS repeat-measurement after the given treatment

DETAILED DESCRIPTION:
SUMMARY

Rationale: In clinical practice the position of TENS electrodes appears to be critical to success. It is claimed that electrodes should target areas with high neural density and where nerve bundles come close to the body surface. These areas are likely to have low skin resistances. Research in the field of electro-analgesia suggests areas of low skin resistance are linked to TENS stimulation points, and that this lower skin resistance may reflect areas with a higher density of neural tissue. When stimulated these areas are likely to generate larger nerve activity and potentially a greater analgesic outcome. For this reason many acupuncturist use a point finder to locate the optimal site to insert the acupuncture needle. To date the relationship between the skin resistance of the areas stimulated by TENS and pain relief is not known.

At present, optimal sites for electrode positioning is made ad hoc using a trial and error approach. This may result in electrodes being positioned at sub-optimal sites. The Philips new electronic pain relief device contains an array, or matrix, of small electrodes. Using this array, the device can measure electrical skin properties. In addition, the user can select which electrodes in the array are active and can adjust the intensity of those electrodes so that stimulation can be targeted to a specific location. In this way it is possible to investigate whether stimulating areas of low skin resistance has an effect on pain relief.

With a novel matrix TENS electrode we would like to investigate the TENS outcome for different electrode specifically chosen locations versus randomly chosen locations. Randomly chosen locations are defined as an area of approximately 10x10 cm around the specifically chosen location in which the random simulation point is chosen. The outcome of the specific vs. random stimulation will be measured with as primary outcome pain and mobility and as secondary outcome strength, joint range, and quality of life.

Objective: Determine effects of transcutaneous electrical nerve stimulation (TENS) on pain and mobility by comparing different stimulation sites; 1) the location with the lowest resistance, 2) the location that causes an irradiation sensation, 3) a random stimulation site (but within a 10x10cm area of the irradiation site). The effect is defined as the pain VAS baseline-measurement before treatment minus the pain VAS repeat-measurement after the given treatment

Study design: double-blind intervention study

Study population: Patients with chronic pain arise from osteo-arthritis in one or both knees Age (>18y), sex and ethnic background are not relevant

Intervention (if applicable): Patients receive a 3 times 30 minutes TENS treatment.

Main study parameters/endpoints: The primary outcome parameters are pain (VAS) and mobility (PDI and 6 min walk). Secondary outcome parameters are strength (MVC) and range-of-motion (ROM) in knee extension and quality of life (SF36).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is no risk for the patients. The burden for the participants is 3 times 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* osteo-arthritis patients diagnosed by medical professional
* at least 18 years old
* VAS higher than 40mm, lower than 70mm (on a 100 mm VAS scale) at the moment of the investigation
* pain symptoms duration longer than 3 months

Exclusion Criteria:

* unable to comprehend instructions
* unable to co-operate
* malignancy
* recent bleeding tissue or haemorrhage in knee
* epilepsy
* advanced cardiovascular conditions, e.g. severe angina or cardiac arrhythmias
* Pacemakers or cochlear implants
* pregnant
* sensory loss of the area to be treated
* devitalised skin e.g. after recent radiotherapy;
* local acute skin conditions e.g. eczema, dermatitis
* doubtful diagnoses
* global, multiple location pain (other than both knees)
* people who undergo currently a TENS treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determine the effect of TENS on pain and mobility for each treatment group separately. Also determine the differences of the effect of TENS by comparing different stimulation sites; | 1 year
  outcomes of the tests are stored at the PC. If all results of all patients are ready. Results will be statistically analysed.This will be in 1 year.

SECONDARY OUTCOMES:
relationship between skin resistance values before stimulation with the sensations during TENS.Explore whether there is a relation between physiological or psychological characteristics of patients and outcome of TENS and user satisfaction questionnaire | 1 year
  outcomes of the tests are stored at the PC. If all results of all patients are ready. Results will be statistically analysed.This will be in 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: A Kolen, PhD, Principal Investigator — Philips Research Eindhoven
Locations (1):
- Maxima Medical Centre, Eindhoven, North Brabant, Netherlands